CLINICAL TRIAL: NCT04243122
Title: A Phase 2 Pilot Randomized Controlled Trial Assessing Feasibility of Thromboprophylaxis With Apixaban in JAK2-positive Myeloproliferative Neoplasm Patients
Brief Title: Assessing Feasibility of Thromboprophylaxis With Apixaban in JAK2-positive Myeloproliferative Neoplasm Patients
Acronym: AIRPORT-MPN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network); the Association médicale universitaire de l'Hôpital Montfort (AMUHM) (Unknown); Canadian Hematology Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AIRPORT-MPN-001
Record Dates: First submitted 2020-01-06; First posted 2020-01-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Myeloproliferative Neoplasm (MPN); Essential Thrombocythemia (ET); JAK2 Mutation; Polycythemia Vera (PV); Primary Myelofibrosis; Venous Thromboembolism (VTE)
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis; Venous Thromboembolism | interventions — apixaban; Tablets; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin and cytoreductive therapy (if applicable) (Active Comparator): Patients who are randomized to this group will take a low-dose aspirin 81mg pill once per day (standard-of-care) for at least 6 months along with cytoreductive therapy, if applicable. Patients will then be treated and followed up as per standard of care at the discretion of his or her treating physician after the completion of the study.
  Interventions: Drug: Aspirin 81 mg
- Apixaban and cytoreductive therapy (if applicable) (Experimental): Patients who are randomized to this group will receive apixaban 2.5mg twice daily for at least 6 months along with standard intervention, cytoreductive therapy, if applicable. Patients will then be treated and followed up as per standard of care at the discretion of their treating physician after the completion of the study.
  Interventions: Drug: Apixaban 2.5 MG Oral Tablet [ELIQUIS]

INTERVENTIONS:
Drug: Apixaban 2.5 MG Oral Tablet [ELIQUIS] — 2.5mg twice per day for 6 months Then treated & followed up as per standard of care
  Other Names: Eliquis
  Arms: Apixaban and cytoreductive therapy (if applicable)
Drug: Aspirin 81 mg — 81mg once per day for 6 months Then treated & followed up as per standard of care
  Other Names: Acetylsalicylic acid
  Arms: Aspirin and cytoreductive therapy (if applicable)

SUMMARY:
Myeloproliferative neoplasms (MPNs) are blood disorders that occur when the body makes too many white or red blood cells, or platelets. This overproduction of blood cells in the bone marrow can create problems for blood flow and lead to various symptoms. One of the major problems is the formation of blood clots. These may form in the veins of a patient's legs or arms where they cause leg or arm pain, swelling or difficulty walking. These clots may travel to the lung and then cause chest pain, shortness of breath and sometimes death. Blood clots can also lead to poor or no blood flow to one's heart, brain, or other organs, causing damages that cannot be easily or ever repaired, such as stroke or heart attack.

Patients diagnosed with certain types of MPN are associated with a higher risk of developing blood clots and related complications. For this reason, MPN patients are usually treated with low-dose aspirin, a common drug used for blood clot prevention, on long-term basis to prevent the formation of blood clots and other complications. However, recent studies also show that the risk of blood clots remains elevated in MPN patients treated with aspirin, and there may not be improvement or reduction in fatal or other events that are associated with blood clots. In addition, since this medical condition is rare, so there's a lack of studies done with high quality results to help physicians decide the best treatment plan for these patients.

The study drug, apixaban, is a new type of orally-taken blood thinner that has been shown to be effective and safe for prevention and treatment of blood clots in various patient populations. The investigators will evaluate whether apixaban is safer and/or better at preventing blood clots and other complications in MPN patients compared to aspirin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older,
2. Confirmed diagnosis of PV, JAK2ET or JAK2 pre-fibrotic MF, per local clinical definitions
3. Able and willing to comply with study procedures and follow-up examinations contained within the written consent form

Exclusion Criteria:

1. Known allergy to apixaban or aspirin,
2. Another need for anticoagulation or specific anti-platelet therapy,
3. Contraindication to thromboprophylaxis (which would specifically include but not be limited to platelets less than 50x10^9/L and acquired Von Willebrand disease),
4. Current pregnancy or breast-feeding,
5. Renal dysfunction (Creatine Clearance <25 mL/min),
6. Known liver disease
7. Currently on any medication with a known interaction to apixaban
8. Unwilling to use an effective means of contraception for women of childbearing potential
9. Overtly fibrotic myelofibrosis
10. Myelodysplastic/myeloproliferative neoplasms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Average monthly subject recruitment rate of all study sites during a 6-month recruitment period | For the duration of study enrollment period: 6 months
Number of JAK2MPN patients recruited in 6 months in comparison to a target recruitment total of 39 prevalent cases and 5 incident cases at minimum | For the duration of study enrollment period: 6 months
Study Feasibility 1: Feasibility of recruitment | For the duration of study enrollment period: 6 months
  Feasibility of recruitment efforts will be determined by the proportion of patients contacted for screening versus those who are consented
Study Feasibility 2: Feasibility of enrollment | For the duration of study enrollment period: 6 months
  Feasibility of enrollment will be determined by the proportion of patients consented vs those were enrolled and randomized
Study Feasibility 3: Patient retention rate | For the duration of the study follow-up period: 7 months
  This will be defined as the proportion of patients who started study intervention versus those who completed each of the study follow-up visits.
Quality of life on apixaban and aspirin will be measured through the use of the RAND 36-Item Health Survey (SF-36), with scores being transformed into a 0-100 scale where the higher the score the less disability. | For the duration of the study follow-up period: 7 months

SECONDARY OUTCOMES:
Study drug compliance as assessed by the proportion of study drug prescribed to the patient versus the actual amount study drug taken by the patient | For the duration of the study follow-up period: 7 months
Study visit compliance as assessed by the number of study visits (in person and/or phone call) completed | For the duration of the study follow-up period: 7 months
Percentage of incident and prevalent cases included in the study | For the duration of study enrollment period: 6 months
Rate of combined arterial and venous thrombotic events (MI, stroke, transient ischemic attack, peripheral arterial thrombosis, VTE) | For the duration of the study follow-up period: 7 months
  This will be defined as the total number of arterial and venous thrombotic events developed relative to the total number of patients who received study treatment
Rate of major bleeding as per the International Society of Thrombosis and Hemostasis definitions | For the duration of the study follow-up period: 7 months
  This will be defined as the total number of adjudicated major bleeding events relative to the total number of patients who received study treatment
Rate of non-major clinically relevant bleeding as per the International Society of Thrombosis and Hemostasis definitions | For the duration of the study follow-up period: 7 months
  This will be defined as the total number of adjudicated non-major clinically relevant bleeding events relative to the total number of patients who received study treatment
Rate of all-cause mortality | For the duration of the study follow-up period: 7 months
  This will be defined as the total number of adjudicated deaths relative to the total number of patients who received study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aurelien Delluc, MD, PhD, Principal Investigator — The Ottawa Hospital; Miriam Kimpton, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No